CLINICAL TRIAL: NCT01679509
Title: Prospective Randomized Comparison of Single-port and Three-port Laparoscopic Adnexal Surgery
Brief Title: Study of Laparoendoscopic Single Site Adnexal Surgery for Benign Ovarian and Tubal Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Joo-Hyun Nam, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LESS-A
Record Dates: First submitted 2012-09-03; First posted 2012-09-06 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Benign Ovarian or Tubal Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single-port surgery group (Experimental): Single-port laparoscopic adnexal surgery
  Interventions: Procedure: Single-port laparoscopic adnexal surgery
- Three-port surgery group (Active Comparator): Three-port laparoscopic adnexal surgery
  Interventions: Procedure: Three-port laparoscopic adnexal surgery

INTERVENTIONS:
Procedure: Single-port laparoscopic adnexal surgery
  Arms: Single-port surgery group
Procedure: Three-port laparoscopic adnexal surgery
  Arms: Three-port surgery group

SUMMARY:
To compare the safety and efficacy between single-port and three-port adnexal surgery in patients with benign ovarian and tubal disease

ELIGIBILITY:
Inclusion Criteria:

* Patient who undergo laparoscopic adnexal surgery due to following benign adenxal disease

  1. Benign teratoma
  2. Endometrioma
  3. Mucinous cystadenoma
  4. Serous cystadenoma
  5. Benign Brenner tumor
  6. Ectopic pregnancy(cornual, tubal, ovarian pregnancy, etc.)
  7. paratubal cyst, parovarian cyst
  8. Risk reducing bilateral salpingooophorecotmy due to familial breast/ovarian cancer syndrome
  9. Other benign adnexal disease requiring surgery
* American Society of Anesthesiologist Physical Status classification I-II.
* Patient who have signed written informed consent

Exclusion Criteria:

* Uncontrolled medical disease
* Active infectious disease
* Previous pelvic radiation therapy
* Patient who requires further procedure excluding adnexal surgery
* Patient who has other pain source excluding adnexal disease
* Pregnant and lactating woman

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2012-09; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
postoperative hospital stay | within 1 week after surgery

SECONDARY OUTCOMES:
postoperative pain | within 1 week after surgery
postoperative analgesics requirement | within 1 week after surgery
quality of life | within 6 months aftr surgery
surgical stress response | within 2 days after surgery
operating time | immediately ater surgery
transfusion requirement and amount | within 1 week after surgery
postoperative complication | within 1 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Hyun Nam, M.D., Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Department of Obstetrics and Gynecology, Universit of Ulsan College of Medicine, Asan Medical Center, Seoul, South Korea